CLINICAL TRIAL: NCT00412061
Title: A Randomized, Double-blind Placebo-controlled, Multicenter Phase III Study in Patients With Advanced Carcinoid Tumor Receiving Octreotide Depot and Everolimus 10 mg/Day or Octreotide Depot and Placebo
Brief Title: Everolimus and Octreotide in Patients With Advanced Carcinoid Tumor
Acronym: RADIANT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRAD001C2325; 2006-004507-18 (EudraCT Number)
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Carcinoid Tumor; Malignant Carcinoid Syndrome
Keywords: Cancer; Carcinoid; Tumor; Neuroendocrine; Carcinoma; Everolimus; Octreotide
MeSH Terms: conditions — Carcinoid Tumor; Malignant Carcinoid Syndrome; Neoplasms; Carcinoma | interventions — Octreotide; Everolimus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Octreotide+ Everolimus (Experimental): Everolimus was administered in accordance with a 10-mg daily dosing regimen (two 5-mg tablets) in conjunction with octreotide 30 mg intramuscularly (i.m.) every 28 days. Patients were treated until progression or unacceptable toxicity. Each treatment cycle lasted 28 days. Patients received their first dose of everolimus at Cycle 1, Day 1. Administration of octreotide was performed every 28 days (± 4 days) starting on Cycle 1, Day 1.
  Interventions: Drug: Octreotide; Drug: Everolimus
- Octreotide+ Placebo (Placebo Comparator): Matching placebo was administered in accordance with a 10-mg daily dosing regimen (two 5-mg tablets) in conjunction with octreotide 30 mg intramuscularly (i.m.) every 28 days. Patients were treated until progression or unacceptable toxicity; Each treatment cycle lasted 28 days. Patients received their first dose of matching placebo at Cycle 1, Day 1. Administration of octreotide was performed every 28 days (± 4 days) starting on Cycle 1 Day 1.
  Interventions: Drug: Octreotide; Drug: Placebo

INTERVENTIONS:
Drug: Octreotide — Octreotide 30 mg intramuscularly (i.m.) every 28 days.
  Other Names: Sandostatin LAR® Depot
Drug: Placebo — A 10-mg oral daily dosing regimen (two 5-mg tablets) of matching placebo.
  Arms: Octreotide+ Placebo
Drug: Everolimus — A 10-mg oral daily dosing regimen (two 5-mg tablets) of everolimus.
  Other Names: RAD001
  Arms: Octreotide+ Everolimus

SUMMARY:
The purpose of this study was to evaluate whether everolimus 10 mg / day added to treatment with depot octreotide prolongs progression free survival compared to treatment with octreotide alone in patients with advanced carcinoid tumor.

ELIGIBILITY:
Inclusion criteria:

* Advanced (unresectable or metastatic) carcinoid tumor
* Confirmed low-grade or intermediate-grade neuroendocrine carcinoma
* Documented progression of disease within 12 months prior to randomization.
* Measurable disease determined by triphasic computer tomography (CT) scan or magnetic resonance imaging (MRI).

Exclusion criteria:

* Poorly differentiated neuroendocrine carcinoma, high-grade neuroendocrine carcinoma, adenocarcinoid, goblet cell carcinoma, or small cell carcinoma.
* Hepatic artery embolization within the last 6 months or cryoablation of hepatic metastasis within 2 months of enrollment.
* Previous treatment with mammalian target of rapamycin (mTOR) inhibitors (sirolimus, temsirolimus, everolimus)
* Intolerance or hypersensitivity to octreotide, everolimus, or other rapamycins.
* Severe or uncontrolled medical conditions
* Chronic treatment with corticosteroids or other immunosuppressive agent.
* Other primary cancer within 3 years.

Other protocol-defined inclusion/exclusion criteria applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2006-12; Primary Completion 2010-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (68):
- United States (38):
  - University of Arizona / Arizona Cancer Center Deptof Uof A/Arizona Cancer(2), Tucson, Arizona
  - Highlands Oncology Group The Center for Chest Care, Fayetteville, Arkansas
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Cedars Sinai Medical Center SC-2, Los Angeles, California
  - University of California at Los Angeles UCLA New SC Address, Los Angeles, California
  - University of Colorado Dept. of Univ. of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Centers Dept of Rocky Mountain (2), Denver, Colorado
  - Eastern Connecticut Hematology & Oncology Associates Dept. of ECHO, Norwich, Connecticut
  - Cancer Centers of Connecticut Southington Location, Southington, Connecticut
  - Hematology Oncology PC Dept.of Hematology Oncology(2), Stamford, Connecticut
  - Ocala Oncology Center Dept. of Ocala Oncology Center, Ocala, Florida
  - Cancer Care and Hematology Specialists of Chicagoland Niles, Niles, Illinois
  - Indiana University Dept.of IndianaUniv.CancerCtr, Indianapolis, Indiana
  - Central Indiana Cancer Centers CICC - South, Indianapolis, Indiana
  - University of Iowa Medical Center Internal Medicine, Iowa City, Iowa
  - University of Kansas Cancer Center Deptof Uof Kansas CancerCenter, Kansas City, Kansas
  - Kansas City Cancer Center KCCC Business Office, Overland Park, Kansas
  - Norton Cancer Institute Clinical Research Program, Louisville, Kentucky
  - LSU HEALTH SCIENCES CENTER/ LSU SCHOOL OF MEDICINE Deptof LSU Health Sciences (2), New Orleans, Louisiana
  - Mayo Clinic - Rochester Division of Hematology, Rochester, Minnesota
  - Washington University School Of Medicine-Siteman Cancer Ctr Division of Oncology, St Louis, Missouri
  - The Center for Cancer Care and Research, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center Medical Oncology, Lebanon, New Hampshire
  - New York Oncology Hematology, P.C. Dept. of New York Oncology. PC, Albany, New York
  - New York University Medical Center NYU Medical Center (2), New York, New York
  - Duke University Medical Center Dept. of Duke Cancer Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas CC of C -Eastside, Greenville, South Carolina
  - Texas Oncology, P.A. Central Austin Cancer Center, Austin, Texas
  - South Texas Institute of Cancer S. Tex Inst.- Corpus Christi, Corpus Christi, Texas
  - Sammons Cancer Center - Texas Oncology Sammons Cancer Center (SC), Dallas, Texas
  - Texas Oncology, P.A. Forth Worth -- 12th Avenue, Fort Worth, Texas
  - University of Texas/MD Anderson Cancer Center Gastrointestinal Med. Oncology, Houston, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates VOA - Lake Wright, Norfolk, Virginia
  - Northwest Cancer Specialists Compass Oncology -BKM, Vancouver, Washington
  - University of Wisconsin / Paul P. Carbone Comp Cancer Center GI Oncology Research Center, Madison, Wisconsin
- Australia (3):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
- Novartis Investigative Site, Brussels, Belgium
- Canada (3):
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (2):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Příbram
- Novartis Investigative Site, Helsinki, Finland
- France (7):
  - Novartis Investigative Site, Strasbourg, France
  - Novartis Investigative Site, Clichy Cédex
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
- Novartis Investigative Site, Athens, Greece, Greece
- Italy (4):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
- Netherlands (2):
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Bratislava, Slovak Republic, Slovakia
- Novartis Investigative Site, Madrid, Madrid, Spain
- Novartis Investigative Site, Uppsala, Sweden
- Novartis Investigative Site, Basingstoke, United Kingdom

REFERENCES:
- [Derived] Pavel ME, Baudin E, Oberg KE, Hainsworth JD, Voi M, Rouyrre N, Peeters M, Gross DJ, Yao JC. Efficacy of everolimus plus octreotide LAR in patients with advanced neuroendocrine tumor and carcinoid syndrome: final overall survival from the randomized, placebo-controlled phase 3 RADIANT-2 study. Ann Oncol. 2017 Jul 1;28(7):1569-1575. doi: 10.1093/annonc/mdx193. PMID 28444114
- [Derived] Fazio N, Granberg D, Grossman A, Saletan S, Klimovsky J, Panneerselvam A, Wolin EM. Everolimus plus octreotide long-acting repeatable in patients with advanced lung neuroendocrine tumors: analysis of the phase 3, randomized, placebo-controlled RADIANT-2 study. Chest. 2013 Apr;143(4):955-962. doi: 10.1378/chest.12-1108. PMID 23187897
- [Derived] Pavel ME, Hainsworth JD, Baudin E, Peeters M, Horsch D, Winkler RE, Klimovsky J, Lebwohl D, Jehl V, Wolin EM, Oberg K, Van Cutsem E, Yao JC; RADIANT-2 Study Group. Everolimus plus octreotide long-acting repeatable for the treatment of advanced neuroendocrine tumours associated with carcinoid syndrome (RADIANT-2): a randomised, placebo-controlled, phase 3 study. Lancet. 2011 Dec 10;378(9808):2005-2012. doi: 10.1016/S0140-6736(11)61742-X. Epub 2011 Nov 25. PMID 22119496
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 429 patients were randomized to double blind phase of treatment. 170 patients moved to the Open Label Phase.
Groups:
- Octreotide+ Placebo Followed by Open Label Arm: Matching placebo was administered in accordance with a 10-mg daily dosing regimen (two 5-mg tablets) in conjunction with octreotide 30 mg intramuscularly (i.m.) every 28 days. Patients were treated until progression or unacceptable toxicity; Each treatment cycle lasted 28 days. Patients received their first dose of matching placebo at Cycle 1, Day 1. Administration of octreotide was performed every 28 days (± 4 days) starting on Cycle 1 Day 1. Open Label - Patients who had progressive disease in this arm, can move to the open label Everolimus + depot octreotide by choice.
Period: Double Blind Phase
Arm/Group | Octreotide+ Everolimus | Octreotide+ Placebo Followed by Open Label Arm
Started | 216 | 213
Safety Set | 215 (1 patient did not provide at laest one valid post baseline safety assessment.) | 211 (1 pt randomized never took drug Another randomized did not have valid post BL safety assessment)
Completed | 0 | 0
Not Completed | 216 | 213
Not completed — Disease Progression | 101 | 154
Not completed — Adverse Event | 61 | 16
Not completed — Final Primary Analysis | 26 | 14
Not completed — Withdrawal by Subject | 18 | 20
Not completed — Death | 6 | 3
Not completed — Protocol Violation | 3 | 4
Not completed — New Cander Therapy | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Open Label Phase
Arm/Group | Octreotide+ Everolimus | Octreotide+ Placebo Followed by Open Label Arm
Started | 0 | 170
Completed | 0 | 0
Not Completed | 0 | 170
Not completed — Disease Progression | 0 | 86
Not completed — Adverse Event | 0 | 46
Not completed — Withdrawal by Subject | 0 | 15
Not completed — Administrative Problems | 0 | 13
Not completed — Death | 0 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — New Cancer Therapy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide+ Everolimus | Octreotide+ Placebo | Total
Number analyzed (Participants) | 216 | 213 | 429
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.72) | 59.4 (11.13) | 59.8 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 89 | 208
  Male | 97 | 124 | 221

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Per Adjudicated Central Radiology Review
Description: Progression free survival (PFS) is defined as the time from randomization to the date of first documented disease progression or death from any cause. The primary analysis of PFS was based on the independent central adjudicated assessment using Kaplan-Meier method.
Time Frame: Time from randomisation to dates of disease progression, death from any cause or last tumor assessment, reported between day of first patient randomised, 10 January 2007, until cut-off date 02 April 2010
Population: The Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Octreotide+ Everolimus | Octreotide+ Placebo
Number analyzed (Participants) | 216 | 213
Months | 16.43 [13.67 to 21.19] | 11.33 [8.44 to 14.59]

2. Secondary Outcome: Best Overall Response Rate as Per Adjudicated Central Radiology Review Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: The best overall response rate is defined as the percentage of patients having achieved confirmed Complete Response + Partial Response. Complete Response (CR) = at least two determinations of CR at least 4 weeks apart before progression. • Partial response (PR) = at least two determinations of PR or better at least 4 weeks apart before progression.
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS; Intent-to-treat Population) consists of all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Octreotide+ Everolimus | Octreotide+ Placebo
Number analyzed (Participants) | 216 | 213
Percentage of patients | 2.3 [0.8 to 5.30] | 1.9 [0.5 to 4.7]

3. Secondary Outcome: Progression Free Survival (PFS) as Per Adjudicated Central Review by Baseline 5-hydroxyindoleacetic Acid (5-HIAA) Level
Description: 5-HIAA levels in urine are frequently elevated in patients with advanced carcinoid tumors. Baseline levels of 5-HIAA in urine were defined as 'High' if they exceeded the median value, and 'Low' if they were lower than or equal to the median.
Time Frame: If elevated at baseline, evaluated every cycle visit (28 days/cycle) reported between day of first patient randomised, 10 January 2007, until cut-off date 02 April 2010
Population: The Full Analysis Set (FAS; Intent-to-treat Population) consists of all randomized patients. This analysis includes PFS patients with non missing baseline 5-HIAA data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Octreotide+ Everolimus | Octreotide+ Placebo
Number analyzed (Participants) | 187 | 191
Months
  5-HIAA <=median (n=93,96) | 21.75 [13.93 to NA] — Upper Limit was not applicable or computable as median was just reached. | 13.90 [8.71 to 22.44]
  5-HIAA > median (n=94,95) | 13.83 [10.61 to 18.63] | 8.41 [8.08 to 11.33]

4. Secondary Outcome: Overall Survival Using Kaplan-Meier Methodology
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause. If a patient was not known to have died, survival was censored at the date of last contact. Kaplan-Meier methodology was used to estimate the median overall survival for each treatment group.
Time Frame: Months 12, 24, 36, 48
Population: The Full Analysis Set (FAS; Intent-to-treat Population) consists of all randomized patients.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Octreotide+ Everolimus | Octreotide+ Placebo Followed by Open Label Arm
Number analyzed (Participants) | 216 | 213
Percentage of Participants
  12 Months | 80.5 [74.5 to 85.3] | 81.8 [75.8 to 86.4]
  24 Months | 57.0 [49.9 to 63.4] | 63.6 [56.6 to 69.8]
  36 Months | 42.9 [36.0 to 49.6] | 48.5 [41.4 to 55.3]
  48 Months | 38.0 [31.2 to 44.7] | 41.6 [34.6 to 48.5]

5. Secondary Outcome: Number of Patients With Adverse Events (AEs), Clinically Notable AE, Death, Serious Adverse Events (SAEs) (Double-Blind Phase)
Description: AEs are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. SAEs are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: From first day of treatment up to 28 days after last day of treatment in double blind
Population: The Safety Set consists of all patients who received at least one dose of study drug and who had at least one valid post-baseline safety assessment.
Measure: Number; unit: Patients
Arm/Group | Octreotide+ Everolimus | Octreotide+ Placebo
Number analyzed (Participants) | 215 | 211
Patients
  Clinically notable AE | 208 | 146
  Grade 3-4 Adverse Events | 162 | 109
  On treatment death | 19 | 11
  Serious adverse events | 126 | 74

6. Secondary Outcome: Number of Patients With Adverse Events (AEs), Clinically Notable AE, Death, Serious Adverse Events (SAEs) (Open Label Phase)
Description: as for outcome 5
Time Frame: From first day of treatment up to 28 days after last day of treatment in double blind
Population: as for outcome 5
Measure: Number; unit: Patients
Groups:
- Everolimus Open Label Arm: Patients who had progressive disease in this arm, can move to the open label Everolimus + depot octreotide by choice.
Arm/Group | Everolimus Open Label Arm
Number analyzed (Participants) | 170
Patients
  Clinically notable AE | 154
  Grade 3-4 Adverse Events | 115
  On treatment death | 22
  Serious adverse events | 93

7. Secondary Outcome: Progression Free Survival (PFS) as Per Adjudicated Central Review by Baseline Chromogranin A (CgA)
Description: Serum CgA levels in urine are frequently elevated in patients with advanced carcinoid tumors. Baseline levels of serum CgA were characterized relative to the upper limited of normal (ULN). CgA levels exceeding 2 x ULN were considered to be 'Elevated'; otherwise considered as "Non-elevated".
Time Frame: as for outcome 3
Population: The Full Analysis Set (FAS; Intent-to-treat Population) consists of all randomized patients. This analysis includes PFS patients with non missing baseline CgA data.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Octreotide+ Everolimus | Octreotide+ Placebo
Number analyzed (Participants) | 212 | 208
Months
  CgA<=2x ULN (n=60,78) | 31.31 [19.32 to NA] — Upper Limit was not applicable or computable as median was just reached. | 20.07 [13.04 to NA] — Upper Limit was not applicable or computable as median was just reached.
  CgA>2x ULN (n=152,130) | 13.93 [11.30 to 17.08] | 8.41 [7.72 to 11.14]

ADVERSE EVENTS:
Description: Double blind period, Safety Set consists all patients received at least one dose of study drug and who had at least one valid post-baseline safety assessment. The Open-label Set consists all patients received at least one dose of open-label everolimus and who had at least one valid safety assessment after initiation of open-label treatment
Groups:
- Everolimus + Octreotide: Everolimus was administered in accordance with a 10-mg daily dosing regimen (two 5-mg tablets) in conjunction with octreotide 30 mg intramuscularly (i.m.) every 28 days. Patients were treated until progression or unacceptable toxicity. Each treatment cycle lasted 28 days. Patients received their first dose of everolimus at Cycle 1, Day 1. Administration of octreotide was performed every 28 days (± 4 days) starting on Cycle 1, Day 1.
- Placebo + Octreotide: Matching placebo was administered in accordance with a 10-mg daily dosing regimen (two 5-mg tablets) in conjunction with octreotide 30 mg intramuscularly (i.m.) every 28 days. Patients were treated until progression or unacceptable toxicity; Each treatment cycle lasted 28 days. Patients received their first dose of matching placebo at Cycle 1, Day 1. Administration of octreotide was performed every 28 days (± 4 days) starting on Cycle 1 Day 1.
- Everolimus Open Label: Open Label - Patients who had progressive disease in this arm, can move to the open label Everolimus + depot octreotide by choice.
Arm/Group | Everolimus + Octreotide | Placebo + Octreotide | Everolimus Open Label
Serious Adverse Events (participants affected / at risk) | 126/215 | 74/211 | 93/170
Other Adverse Events (participants affected / at risk) | 214/215 | 194/211 | 162/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Octreotide (N=215) | Placebo + Octreotide (N=211) | Everolimus Open Label (N=170)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 3 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Carcinoid heart disease (Cardiac disorders) | 2 | 2 | 2
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 2 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Dilatation ventricular (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Mitral valve stenosis (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pulmonary valve incompetence (Cardiac disorders) | 0 | 1 | 0
Pulmonary valve stenosis (Cardiac disorders) | 1 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0
Tricuspid valve disease (Cardiac disorders) | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 2 | 0
Tricuspid valve prolapse (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve stenosis (Cardiac disorders) | 0 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0
Carcinoid crisis (Endocrine disorders) | 1 | 0 | 1
Carcinoid syndrome (Endocrine disorders) | 2 | 1 | 2
Diplopia (Eye disorders) | 0 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 15 | 11 | 11
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1
Ascites (Gastrointestinal disorders) | 0 | 5 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 5 | 7
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 5 | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal angina (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 5 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 2
Lip oedema (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 4 | 4 | 2
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 8 | 3 | 4
Small intestinal stenosis (Gastrointestinal disorders) | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Subileus (Gastrointestinal disorders) | 3 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 6 | 5
Asthenia (General disorders) | 2 | 3 | 1
Brain death (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 1
Chills (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 0
General physical health deterioration (General disorders) | 6 | 3 | 5
Generalised oedema (General disorders) | 1 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 2 | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 0 | 0
Oedema peripheral (General disorders) | 3 | 4 | 3
Pain (General disorders) | 1 | 2 | 0
Performance status decreased (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 8 | 3 | 3
Spinal pain (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 1
Abscess intestinal (Infections and infestations) | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0
Aspergillosis (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 3 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 2
Lung infection (Infections and infestations) | 1 | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 9 | 1 | 5
Pneumonia viral (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 4
Sinusitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 4
Blood urea increased (Investigations) | 1 | 0 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0
Coagulation time shortened (Investigations) | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 7 | 1 | 3
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
B-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung infiltration malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Intracranial haematoma (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 2
Confusional state (Psychiatric disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Bladder tamponade (Renal and urinary disorders) | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0
Eosinophilic cystitis (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 2
Renal failure (Renal and urinary disorders) | 4 | 0 | 3
Renal failure acute (Renal and urinary disorders) | 3 | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1
Renal infarct (Renal and urinary disorders) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 1
Granulomatous pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 2
Flushing (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus + Octreotide (N=215) | Placebo + Octreotide (N=211) | Everolimus Open Label (N=170)
Anaemia (Blood and lymphatic system disorders) | 58 | 21 | 34
Leukopenia (Blood and lymphatic system disorders) | 16 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 18 | 3 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 34 | 1 | 15
Abdominal distension (Gastrointestinal disorders) | 12 | 12 | 10
Abdominal pain (Gastrointestinal disorders) | 65 | 68 | 43
Abdominal pain upper (Gastrointestinal disorders) | 22 | 26 | 16
Aphthous stomatitis (Gastrointestinal disorders) | 28 | 3 | 15
Ascites (Gastrointestinal disorders) | 17 | 9 | 8
Constipation (Gastrointestinal disorders) | 31 | 22 | 17
Diarrhoea (Gastrointestinal disorders) | 114 | 77 | 77
Dry mouth (Gastrointestinal disorders) | 22 | 6 | 7
Dysphagia (Gastrointestinal disorders) | 15 | 5 | 4
Flatulence (Gastrointestinal disorders) | 27 | 28 | 12
Haemorrhoids (Gastrointestinal disorders) | 17 | 9 | 9
Mouth ulceration (Gastrointestinal disorders) | 17 | 5 | 11
Nausea (Gastrointestinal disorders) | 92 | 63 | 60
Stomatitis (Gastrointestinal disorders) | 109 | 25 | 63
Vomiting (Gastrointestinal disorders) | 69 | 40 | 30
Asthenia (General disorders) | 51 | 30 | 30
Chills (General disorders) | 15 | 10 | 5
Fatigue (General disorders) | 103 | 91 | 63
Oedema peripheral (General disorders) | 92 | 47 | 62
Pyrexia (General disorders) | 42 | 21 | 32
Bronchitis (Infections and infestations) | 11 | 7 | 8
Nasopharyngitis (Infections and infestations) | 19 | 26 | 19
Sinusitis (Infections and infestations) | 12 | 9 | 17
Upper respiratory tract infection (Infections and infestations) | 27 | 12 | 11
Urinary tract infection (Infections and infestations) | 27 | 16 | 19
Alanine aminotransferase increased (Investigations) | 9 | 6 | 10
Aspartate aminotransferase increased (Investigations) | 11 | 8 | 8
Blood creatinine increased (Investigations) | 15 | 5 | 8
Weight decreased (Investigations) | 59 | 31 | 33
Decreased appetite (Metabolism and nutrition disorders) | 64 | 36 | 33
Dehydration (Metabolism and nutrition disorders) | 17 | 12 | 9
Hypercholesterolaemia (Metabolism and nutrition disorders) | 17 | 6 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 42 | 9 | 24
Hyperlipidaemia (Metabolism and nutrition disorders) | 15 | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 17 | 4 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 50 | 8 | 27
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 | 5 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 11 | 6 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 28 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 41 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 13 | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 18 | 7 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 21 | 21 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 14 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32 | 24 | 19
Dizziness (Nervous system disorders) | 29 | 24 | 12
Dysgeusia (Nervous system disorders) | 42 | 12 | 30
Headache (Nervous system disorders) | 65 | 49 | 32
Anxiety (Psychiatric disorders) | 14 | 14 | 12
Depression (Psychiatric disorders) | 16 | 11 | 12
Insomnia (Psychiatric disorders) | 20 | 15 | 12
Dysuria (Renal and urinary disorders) | 12 | 5 | 7
Pollakiuria (Renal and urinary disorders) | 10 | 6 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 59 | 32 | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 59 | 19 | 27
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 | 11 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33 | 5 | 24
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 6 | 13
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 6 | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 20 | 2 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 4 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 23 | 5 | 9
Erythema (Skin and subcutaneous tissue disorders) | 17 | 4 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 13 | 5
Onychoclasis (Skin and subcutaneous tissue disorders) | 11 | 1 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 42 | 12 | 18
Rash (Skin and subcutaneous tissue disorders) | 88 | 37 | 59
Flushing (Vascular disorders) | 20 | 20 | 6
Hypertension (Vascular disorders) | 24 | 21 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.